CLINICAL TRIAL: NCT06345183
Title: Real-World Treatment Patterns and Outcomes of Advanced Renal Cell Carcinoma (aRCC) Patients Receiving Nivolumab+Ipilimumab or Pembrolizumab+Lenvatinib in U.S. Oncology Practice
Brief Title: Real-World Outcomes of Nivolumab+Ipilimumab and Pembrolizumab+Lenvatinib Among US Advanced Renal Cell Carcinoma (aRCC) Patients
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-1275
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Advanced Renal Cell Carcinoma (aRCC)
MeSH Terms: interventions — Nivolumab; pembrolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants treated with Nivolumab + Ipilimumab combination therapy
  Interventions: Combination Product: Nivolumab + Ipilimumab combination therapy
- Participants treated with Pembrolizumab + Lenvatinib combination therapy
  Interventions: Combination Product: Pembrolizumab + Lenvatinib combination therapy

INTERVENTIONS:
Combination Product: Nivolumab + Ipilimumab combination therapy — As per product label
  Groups: Participants treated with Nivolumab + Ipilimumab combination therapy
Combination Product: Pembrolizumab + Lenvatinib combination therapy — As per product label
  Groups: Participants treated with Pembrolizumab + Lenvatinib combination therapy

SUMMARY:
This observational study aims to describe demographic, clinical characteristics, treatment patterns outcomes of participants with advanced Renal Cell Carcinoma (aRCC) receiving either Nivolumab + Ipilimumab, or Pembrolizumab + Lenvatinib combination therapy

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older with diagnosis of Advanced Renal Cell Carcinoma (aRCC) with predominantly clear-cell histology
2. Received any of the following therapies in the first-line setting:

   1. Nivolumab + Ipilimumab between 8/1/2021 and 6 months prior to data collection
   2. Pembrolizumab + Lenvatinib between 8/1/2021and 6 months prior to data collection
3. Participant had at least 6 months of follow-up from initiation of index treatment (patients who deceased prior to 6 months since index treatment initiation would still be eligible)

Exclusion Criteria:

1. Receipt of any immunotherapy or tyrosine kinase inhibitor (TKI) therapy as part of a Randomized Controlled Trial (RCT)
2. Participant received any systemic therapy for Advanced Renal Cell Carcinoma (aRCC) prior to index therapy, including neoadjuvant or adjuvant therapy
3. Any active malignancy in the 3 years prior to initiation of 1L therapy for aRCC, except for locally curable cancers that have been cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix, or breast cancer, or localized prostate cancer with a Gleason score ≤3+4 that has been treated more than 12 months prior to full study screening and considered to have a very low risk of recurrence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants diagnosed with advanced Renal Cell Carcinoma (aRCC) who received Nivolumab+Ipilimumab or Pembrolizumab+Lenvatinib combination therapy in the first line (1L) setting
Sampling Method: Non-Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Participant year of birth | Baseline
Participant sex at birth | Baseline
Participant primary payer | Baseline
Participant race | Baseline
Participant ethnicity | Baseline
Participant U.S. state of residence | Baseline
Participant initial Renal Cell Carcinoma (RCC) diagnoses | Baseline
American Joint Committee on Cancer (AJCC) TNM stage | Baseline
Participant advanced/metastatic Renal Cell Carcinoma (RCC) diagnosis | Baseline
Participant renal cell carcinoma (RCC) histology results | Baseline
Participant tumor grade | Baseline
Participant biomarker or genetic testing method | Baseline
Participant molecular and/or genetic mutations reported | Baseline
Participant site of metastatic disease | Index date
Participant Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) | Baseline
Participant Karnofsky score (KPS) | Baseline
Participant comorbidities and/or chronic conditions | Baseline
Participant blood test results | Index date
Participant Memorial Sloan Kettering Cancer Center (MSKCC) score | Index date
Participant International Metastatic Renal-Cell Carcinoma Database Consortium (IMDC) score | index date
Participant smoking status | Baseline
Participant COVID-19 status | Baseline
Participant surgical history | Baseline
Participant radiation treatment history | Baseline
Participant treatment regimen received | Index date up to 32 months
Participant treatment initiation and discontinuation dates | Index date up to 32 months
Participant rationale for discontinuation of treatment | Index date up to 32 months
Participant radiation therapy prescribed | Index date up to 32 months
Participant total number of radiotherapy cycles | Index date up to 32 months
Participant initial dose and frequency/schedule of index therapy | Index date up to 32 months
Participant index treatment dose modifications | Index date up to 32 months
Participant rationale for dose modifications of index therapy | Index date up to 32 months
Participant date of dose modifications of index therapy | Index date up to 32 months
Participant last dose and frequency/schedule of index therapy | Index date up to 32 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Cardinal Health, Dublin, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts